CLINICAL TRIAL: NCT02626806
Title: Exercise-induced High-sensitivity Troponin Levels as a Predictor for Obstructive Coronary Artery Disease
Acronym: EUROCAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Walter Desmet, Head of Clinic, Interventional Cardiology, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: UZL9281
Record Dates: First submitted 2014-04-01; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: exercise test; HS -troponin; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with hemodynamic significant CAD;
- patients without hemodynamic significant CAD

SUMMARY:
1. To compare hs-TnT levels after a cardiac stress test in patients with vs. patients without CAD
2. To assess the level of post-exercise hs-TnT predicting CAD (using ROC-analysis)
3. To determine the sensitivity, specificity and accuracy of this exercise-induced hsTopT level in predicting CAD, either alone or in relation to traditional patient-related and exercise test-related metrics

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected CAD, planned for diagnostic coronary angiogram
2. Patients with previous revascularization, suspected of recurrent ischemia

Exclusion Criteria:

1. Congestive cardiomyopathy with LV EF < 35%
2. Renal failure with eGFR < 30 ml/min
3. Known structural or severe valvular heart disease
4. Prior CABG
5. Previous ACS < 6 weeks
6. Known incomplete revascularization after previous PCI
7. Unstable angina or ACS (defined as unstable anginal symptoms + ECG changes or hs-TnT > 0.053 ng/L)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To compare hs-TnT levels after a cardiac stress test in patients with vs. patients without CAD
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Presence of coronary artery stenosis more than 50% | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium